CLINICAL TRIAL: NCT01029691
Title: Use of PAP in Women With Pre-eclampsia
Brief Title: Study of Positive Airway Pressure in Preeclampsia to Reduce Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Louise O'Brien, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F022873; 1K23HL095739-01 (NIH)
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Preeclampsia; Hypertension
Keywords: Sleep disordered breathing; Preeclampsia; Positive Airway Pressure
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (3):
- Positive Airway Pressure (compliant) (Experimental): This arm was women who used auto-titrating positive airway pressure (APAP) for at least 4 hours per night
  Interventions: Device: Positive Airway Pressure
- Standard care (No Intervention)
- Positive Airway Pressure (non-compliant) (Experimental): No one was assigned to this arm, but for results data quality purposes, women assigned to PAP who were explicitly non-compliant (used less than 4 hours per night), were analyzed separately from women who were compliant with the PAP assignment.
  Interventions: Device: Positive Airway Pressure

INTERVENTIONS:
Device: Positive Airway Pressure — Women will use positive airway pressure until delivery
  Other Names: PAP
  Arms: Positive Airway Pressure (compliant); Positive Airway Pressure (non-compliant)

SUMMARY:
The purpose of this study is to identify whether sleep-disordered breathing - as measured by overnight polysomnography - is associated with pre-eclampsia and to determine whether use of positive airway pressure can improve nocturnal blood pressure.

DETAILED DESCRIPTION:
Initial enrollment began with only women with a pre-existing diagnosis of pre-eclampsia. Part way through the study, IRB granted approval to expand recruitment to include other hypertensive diagnoses. So, in effect, a more accurate post hoc title would be Study of Positive Airway Pressure to Reduce Blood Pressure in Hypertensive Pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Women with preeclampsia who receive care at the University of Michigan Hospitals
* No current use of PAP therapy.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Current PAP therapy
* Any medical reason why PAP therapy may not be suitable (e.g., in patients with recent head trauma).
* Cognitively impaired and unable to understand informed consent.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] O'Brien LM, Bullough AS, Chames MC, Shelgikar AV, Armitage R, Guilleminualt C, Sullivan CE, Johnson TR, Chervin RD. Hypertension, snoring, and obstructive sleep apnoea during pregnancy: a cohort study. BJOG. 2014 Dec;121(13):1685-93. doi: 10.1111/1471-0528.12885. Epub 2014 May 30. PMID 24888772

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women with hypertension were recruited from University of Michigan obstetric clinics and inpatient areas. Enrollment into the trial occurred between March 2010 and November 2013.
Pre-assignment Details: After signing consent, one participant decided not to have any sleep studies performed, explaining the difference between the 125 enrolled listed in the registration section and the 124 followed below.
Groups:
- Compliant Users APAP: Women who used APAP at least 4 hours per night. Auto-titrating Positive Airway Pressure: Women will use APAP until delivery. Nocturnal blood pressure will be assessed at two time points: 1 week of APAP use and at regular intervals across pregnancy. Daytime blood pressure measurements across pregnancy will be obtained from medical records along with delivery information.
- Non-Compliant APAP: Women who were in the APAP arm but who used less than 4 hours per night
- Standard of Care: Women in the standard of care group will have clinical blood pressure measurements extracted from medical records. Delivery information will also be collected.
Period: APAP Initiation to Week 1 or Delivery
Arm/Group | Compliant Users APAP | Non-Compliant APAP | Standard of Care
Started (Assignment to APAP or Standard, not actual beginning of use of APAP vs. standard of care) | 20 | 27 (4 delivered before APAP initiation 7 elected not to have APAP following baseline study) | 77
Baseline Sleep Study | 20 | 23 | 77
Began Actual APAP Use | 20 | 16 | 77
Completed (Women in APAP arm who reached the 1 week blood pressure measure) | 20 | 16 | 77
Not Completed | 0 | 11 | 0
Period: Continued APAP to Delivery
Arm/Group | Compliant Users APAP | Non-Compliant APAP | Standard of Care
Started | 20 | 16 | 77
Completed | 20 | 16 | 76
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: These data are for those who initiated APAP only and do not include the standard of care arm as they did not have nocturnal blood pressure
Groups:
- Compliant Autotitrating Positive Airway Pressure (APAP): Women who used APAP for at least 4 hours/night
- Non-compliant APAP: Women who did not use APAP for at least 4 hours/night
- Standard Care: Non-APAP arm
- Total: Total of all reporting groups
Arm/Group | Compliant Autotitrating Positive Airway Pressure (APAP) | Non-compliant APAP | Standard Care | Total
Number analyzed (Participants) | 20 | 16 | 77 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (4.8) | 32.3 (3.8) | 31.1 (6.6) | 31.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 77 | 113
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 6 | 8 | 19 | 33
  Caucasian | 14 | 6 | 52 | 72
  Asian | 0 | 0 | 2 | 2
  Mixed Race | 0 | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 77 | 113
Nocturnal blood pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 126.7 (9.5) | 124.5 (8.9) | NA (NA) — Standard of care group did not have nocturnal blood pressure measures | 125.8 (9.3)
  Diastolic | 69.7 (8.0) | 68.8 (8.3) | NA (NA) — Standard of care group did not have nocturnal blood pressure measures | 69.3 (8.2)
sleep study apnea hypopnea index (AHI) [Mean (Standard Deviation); unit: events per hour] — Number of respiratory events per hour of sleep
  events per hour | 18.9 (30.6) | 4.2 (6.0) | NA (NA) — The standard of care arm did not undergo a sleep study | 12.4 (24.0)

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Blood Pressure
Description: measured by a 24 hour cuff, averaged across the night;
Time Frame: baseline and 1 week after PAP treatment.
Population: The standard of care group did not have nocturnal blood pressure monitoring as they were not assigned to use a positive airway pressure device
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Positive Airway Pressure Adherent: Positive Airway Pressure: Women will use positive airway pressure until delivery
- Positive Airway Pressure Non Adherent: Positive Airway Pressure: Women who used positive airway pressure for limited time
Arm/Group | Positive Airway Pressure Adherent | Positive Airway Pressure Non Adherent | Standard Care
Number analyzed (Participants) | 20 | 16 | 0
mmHg
  Baseline Nocturnal Systolic | 128.2 (9.8) | 124.7 (8.9) |
  Baseline Nocturnal Diastolic | 70.6 (8.0) | 68.8 (8.3) |
  1 week Systolic: number analyzed (Participants) | 19 | 14 | 0
  1 week Systolic | 127.7 (9.3) | 125.3 (8.5) |
  1 week Diastolic: number analyzed (Participants) | 19 | 14 | 0
  1 week Diastolic | 70.9 (8.4) | 69.3 (7.4) |
Statistical Analysis 1: Comparison: Positive Airway Pressure Adherent vs Positive Airway Pressure Non Adherent vs Standard Care; unadjusted systolic blood pressure at baseline between groups; Test type: Superiority; p = 0.45, t-test, 2 sided
Statistical Analysis 2: Comparison: Positive Airway Pressure Adherent vs Positive Airway Pressure Non Adherent vs Standard Care; Unadjusted diastolic blood pressure at baseline between groups; Test type: Superiority; p = 0.66, t-test, 2 sided
Statistical Analysis 3: Comparison: Positive Airway Pressure Adherent vs Positive Airway Pressure Non Adherent vs Standard Care; Unadjusted systolic blood pressure at week 1; Test type: Superiority; p = 0.61, t-test, 2 sided
Statistical Analysis 4: Comparison: Positive Airway Pressure Adherent vs Positive Airway Pressure Non Adherent vs Standard Care; Unadjusted diastolic blood pressure at week 1; Test type: Superiority; p = 0.75, t-test, 2 sided

2. Primary Outcome: Number of Participants With Worsening of Hypertension
Description: This outcome measure's purpose was to look at the impact of the APAP on blood pressure. This was done categorically by looking at worsening of hypertension with or without escalation of antihypertensive medications.
Time Frame: 1-6 months after enrollment.
Population: One woman in the standard of care group died during pregnancy and is therefore not included in this analysis.
Measure: Number; unit: participants
Arm/Group | Positive Airway Pressure Adherent | Positive Airway Pressure Non Adherent | Standard Care
Number analyzed (Participants) | 20 | 16 | 76
participants | 11 | 9 | 57
Statistical Analysis 1: Comparison: Positive Airway Pressure Adherent vs Positive Airway Pressure Non Adherent vs Standard Care; Test type: Superiority; p = 0.085, Chi-squared

3. Primary Outcome: Severity of Sleep Disordered Breathing
Description: Severity of sleep disordered breathing, using the apnea/hypopnea index (number of respiratory evens per hour of sleep), among participants who have or do not have nocturnal hypertension. Obstructive sleep apnea is typically considered present if the AHI is at least 5.
Time Frame: at baseline
Population: This reflects only the n=43 women who underwent baseline sleep study (n=7 of whom did not go on to receive APAP therapy) prior to assignment to PAP therapy. The standard of care group did not have a baseline sleep study and are therefore not represented here. Of these n=43 women, n=36 received PAP therapy (n=20 were adherent and n=16 were not).
Measure: Mean (Standard Deviation); unit: apnea/hypopnea index
Groups:
- Nocturnal Hypertension: Women with nocturnal hypertension (defined as blood pressure >117/68mmHg between 26-30 weeks and >123/72mmHg after 30 weeks)
- No Nocturnal Hypertension: Women without nocturnal hypertension
Arm/Group | Nocturnal Hypertension | No Nocturnal Hypertension
Number analyzed (Participants) | 29 | 14
apnea/hypopnea index | 15.6 (25.9) | 2.7 (1.9)
Statistical Analysis 1: Comparison: Nocturnal Hypertension vs No Nocturnal Hypertension; Test type: Superiority; p = 0.012, t-test, 2 sided — Unadjusted

4. Primary Outcome: Number of Participants With Sleep-disordered Breathing (SDB)
Description: Presence or absence of SDB (defined as an apnea/hypopnea index; AHI>=5)
Time Frame: Baseline night 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nocturnal Hypertension | No Nocturnal Hypertension
Number analyzed (Participants) | 29 | 14
Participants | 14 | 3

5. Secondary Outcome: Gestational Age at Delivery
Time Frame: At delivery (within 6 months of enrollment).
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Positive Airway Pressure Adherent | Positive Airway Pressure Non Adherent | Standard Care
Number analyzed (Participants) | 20 | 16 | 75
weeks | 36.7 (3.7) | 36.0 (3.6) | 36.9 (3.0)

6. Secondary Outcome: Birth Weight
Time Frame: At delivery (within 6 months of enrollment)
Population: There is one extra baby in each arm to represent the twins born in each group.
Measure: Mean (Standard Deviation); unit: grams
Units Other Than Participants: babies
Arm/Group | Positive Airway Pressure Adherent | Positive Airway Pressure Non Adherent | Standard Care
Number analyzed (Participants) | 20 | 16 | 75
Number analyzed (babies) | 21 | 17 | 76
grams | 2804.3 (1037.4) | 2749.7 (870.0) | 2957.5 (909.3)

7. Secondary Outcome: NICU Admission
Description: Number of mothers who had one (or more) babies admitted to NICU
Time Frame: at delivery (within 6 months of enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Airway Pressure Adherent | Positive Airway Pressure Non Adherent | Standard Care
Number analyzed (Participants) | 20 | 16 | 75
Participants | 1 | 3 | 13
Statistical Analysis 1: Comparison: Positive Airway Pressure Adherent vs Positive Airway Pressure Non Adherent vs Standard Care; Test type: Superiority; p = 0.4, Fisher Exact

ADVERSE EVENTS:
Time Frame: from start of intervention until 30 days after intervention (generally 30 days after delivery)
Description: NOTE: All cause mortality table reflects maternal death only - as babies were not participants.
  Inpatient hospitalizations were not collected as data for adverse event collection (and therefore are not included in Serious Adverse Events reporting) because this was a study of high risk pregnancies, so recruitment came from inpatient candidates as well as from the community.
  For non-serious adverse events: study did not collect ordinary aspects of pregnancy such as nausea.
Arm/Group | Positive Airway Pressure | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/77
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/77
Other Adverse Events (participants affected / at risk) | 0/36 | 0/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Positive Airway Pressure (N=36) | Standard Care (N=77)
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 2 | 0 — pre-existing severe fetal growth restrictions involved in both cases; IRB approved determination that these are unrelated to study participation or intervention. Neonatal deaths not tracked in standard of care arm
medical abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — severe growth restriction of fetus with no interval growth on serial ultrasounds as well as oligohydramnios

LIMITATIONS AND CAVEATS:
These tables represent full basic analysis of all the participants enrolled without adjustment for confounding variables. Future publications will present more complex subsequent analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes